# A NON-RANDOMIZED, CONSECUTIVE ENROLLMENT EVALUATION OF THE DESolve® NOVOLIMUS ELUTING BIORESORBABLE CORONARY SCAFFOLD SYSTEM IN THE TREATMENT OF PATIENTS WITH *DE NOVO* NATIVE CORONARY ARTERY LESIONS

Elixir Medical Clinical Evaluation of the DESolve® Novolimus Eluting Bioresorbable Coronary Scaffold System

"DESolve Nx Trial - DESolve CX Arm"

Revision E, 5 February 2018

**Brazil** 

NCT04034121

#### **CLINICAL STUDY SUMMARY**

| Trial Name and<br>Number | DESolve Nx Trial: ELX-CL-1003 |
|---|---|
| Objectives: | To evaluate the safety, performance and efficacy of the Elixir DESolve® Novolimus Eluting Bioresorbable Coronary Scaffold System (BCSS) in patients with a single <i>de novo</i> native coronary artery lesion designated the target lesion and up to one non-target lesion located in a separate epicardial vessel. |
| Enrollment: | The study is designed to enroll 120 non-randomized patients with a single <i>de novo</i> native coronary artery lesion designated the target lesion and up to one non-target lesion located in a separate epicardial vessel. The target lesion must measure between 2.75 mm and 3.5 mm in diameter and $\leq 10$ mm or $\leq 14$ mm in length able to be covered by a single 3.0 x 14, 3.0 x 18mm, 3.25 x 14 or 3.25 x 18 mm, 3.5 x 14 mm or 3.5 x 18 mm DESolve scaffold. As applicable, a non-target lesion located in a separate epicardial vessel must be treated first with a single, approved 'olimus drug eluting stent and if this procedure is uncomplicated and considered optimal, then the target lesion can be considered for the DESolve Novolimus Eluting BCSS. The patient should not be enrolled until after satisfactory pre-dilatation of the target lesion. Enrollment and follow-up is complete. |
| | The Low Profile 1 study arm is designed to enroll 100 non-randomized patients with a single <i>de novo</i> native coronary artery lesion designated the target lesion and up to one non-target lesion located in a separate epicardial vessel. The target lesion must measure between 2.75 mm and 3.5 mm in diameter and $\leq 10$ mm or $\leq 24$ mm in length able to be covered by a single 3.0, 3.25 or 3.5 mm x 14, 18 or 28 mm scaffold. This device differs only in the thickness of the scaffold which is now 100-120 $\mu$ m as compared to the 150 $\mu$ m of the device previously studied and shown safe and effective. As applicable, a non-target lesion located in a separate epicardial vessel must be treated first with a single, approved 'olimus drug eluting stent and if this procedure is uncomplicated and considered optimal, then the target lesion can be considered for the DESolve Novolimus Eluting BCSS. The patient should not be enrolled until after satisfactory pre-dilatation of the target lesion. Patients included in this |

| | Arm will be enrolled at select sites. Follow-up will conclude at the end of 3 years. |
|---|---|
| Clinical Study Device | 3.0 x 14 mm, 3.0 x 18 mm, and 3.0 x 28mm; 3.25 x 14 mm, 3.25 x 18 mm and 3.25 x 28 mm; 3.5 x 14mm, 3.5 x 18 mm and 3.5 x 28 mm DESolve scaffolds All DESolve scaffolds are loaded with approximately 5 mcg of Novolimus per mm of scaffold length (i.e, 65 mcg on a 14 mm scaffold, 85 mcg on an 18 mm scaffold and 125 mcg on a 28 mm scaffold). |
| Clinical Site<br>Locations: | Drawn from up to 15 International Sites in Brazil, Belgium, Denmark, Germany, Poland and New Zealand |
| Clinical Study Design | The DESolve Nx Trial is a prospective, consecutive enrolment non-randomized study designed to enroll patients with a de novo lesion ≤ 14 mm in length, designated the target lesion, located in a native coronary artery with a reference vessel diameter of 2.75 mm − 3.5 mm. All patients will receive a 3.0, 3.25 or 3.5 mm x 14, 18 or 28 mm scaffold. DESolve scaffold loaded with approximately 5 mcg of Novolimus per mm of scaffold length. As appropriate, a non-target lesion may be treated in a separate native epicardial vessel with a single, approved 'olimus drug eluting stent. Only the target vessel will be evaluated for the key safety and efficacy endpoints. Multiple registry arms are to be included in the study with patients to be enrolled at select sites: |
| | <ul> <li>Low Profile 1 – a lower profile (thinner) scaffold (100-120μm) with the same drug dose</li> </ul> |
| | To provide an assessment of the lesion and scaffold morphology and scaffold strut composition over time, the following additional imaging modalities will be included: |
| | <ul> <li>Angiography will be completed at 6 months following the index<br/>procedure in all patients.</li> </ul> |
| | • In a subset of the first 35 patients enrolled at select sites, IVUS and OCT will be conducted at 6 and 24 and/or 36 months following the index procedure. These patients will also undergo angiography during the 24 and/or 36 month follow-up. |

### Multislice computed tomography (MSCT) will be conducted at 12 months in the subset of the first 35 patients enrolled at select sites. All main trial patients will undergo clinical follow-up at 1, 6, and 12 months and annually through 5 years. LP1 patients will undergo clinical follow-up at 1, 6, and 12 months and annually through 3 years **Clinical Endpoints:** Clinically-indicated Major Adverse Cardiac Events (MACE) at 1, 6, and 12 months and annually to 5 years for all main study patients and for Low Profile 1 (LP1) patients at 1, 6, and 12 months and annually through 3 years. MACE is a composite endpoint defined as cardiac death, target vessel MI, and clinicallyindicated target lesion revascularization Acute Success including Device and Procedure Success Clinically-indicated Target Lesion and Target Vessel Revascularization (CI-TLR and CI-TVR) at 1, 6, and 12 months and annually to 5 years for all main study patients and for LP1 patients at 1, 6, and 12 months and annually through 3 years Clinically-indicated Target Lesion and Target Vessel Failure (CI-TLF and CI-TVF) at 1, 6, and 12 months and annually to 5 years for all main study patients and for LP1 patients at 1, 6, and 12 months and annually through 3 years Scaffold Thrombosis at 1, 6, and 12 months and annually to 5 years for all main study patients and for LP1 patients at 1, 6, and 12 months and annually through 3 years Angiographic All patients will undergo angiographic follow-up at 6 months. In a subset of the first 35 patients enrolled at select sites angiography will also be **Endpoints:** conducted at 24 and/or 36 months. The following endpoints will be analyzed:

In-scaffold late lumen loss

In-lesion Late Lumen Loss

In-scaffold and in-lesion Binary Restenosis (≥ 50%)

| | . I |
|---|---|
| | In-scaffold and in-segment % Diameter Stenosis |
| | MLD and % DS post procedure |
| | Scaffold Thrombosis |
| | Additional parameters may be assessed |
| IVUS and OCT<br>Endpoints | To provide an assessment of the lesion and stent morphology and stent strut composition over time, the additional imaging modalities of IVUS and OCT conducted at baseline, 6 and 24 and/or 36 months will be completed in a subset of the first 35 patients enrolled at select sites. The following endpoints will be analyzed: |
| | Volumetric neointimal burden by IVUS |
| | Changes in vessel size by IVUS |
| | Changes in scaffold size by IVUS |
| | Changes in strut appearance suggesting bioresorption |
| | <ul> <li>Incomplete scaffold apposition, acute and late, assessed by IVUS<br/>and/or Optical Coherence Tomography (OCT)</li> </ul> |
| | Scaffold area assessed by IVUS and/or OCT |
| | Descriptive analysis of lesion/vessel morphormetry and scaffold<br>strut composition by OCT |
| MSCT | In a subset of the first 35 patients enrolled at select sites, MSCT follow-up |
| Analysis Endpoint | will be conducted at 12 months. The following endpoints will be analyzed: |
| | Multi-slice computed tomography (MSCT) descriptive and quantitative analysis of lesion/vessel and scaffold morphology |
| Treatment Strategy | Treatment of up to two de novo native coronary artery lesions located in separate epicardial territories. One will be the target lesion and will be treated with the trial device. |

- Treatment of the target lesion is to be performed after optimal stenting using an approved 'olimus DES of a single non-target lesion as applicable.
- To determine patient eligibility, assessment of the target vessel diameter using on-line QCA must be completed before the enrollment of the patient into the study. The target lesion is to be treated only after all clinical and angiographic inclusion criteria have been met
- Pre-dilatation of the lesion is mandatory using a balloon approximately sized to the reference vessel. If the lesion cannot be successfully pre-dilated, treatment with the DESolve CSS should not be attempted. If there is Type A dissection that cannot be covered by the DESolve CSS then the patient cannot be enrolled in the trial. Any dissection worse than Type A will preclude the patient from being enrolled into the study.
- Target lesion length should be ≤ 10 mm or ≤ 24 mm by visual estimate and have at least 2 mm of healthy vessel on either side of the lesion for coverage by the DESolve Scaffold

Table 1: Lesion length, Scaffold size and Drug dose

| Lesion length (visual estimation) | DESolve Stent size | Drug dose |
|---|---|---|
| ≤ 10 mm | 3.0 x 14 mm<br>3.25 x 14 mm<br>3.5 x 14 mm | 65 mcg |
| ≤ 14 mm | 3.0 x 18 mm<br>3.25 x 18 mm<br>3.5 x 18 mm | 85 mcg |
| ≤ 24 mm | 3.0 x 28 mm<br>3.25 x 28 mm<br>3.5 x 28 mm | 125 mcg |

- Bailout stenting should be conducted using any approved DES stent incorporating an "olimus" drug or bare metal stent
- Patients should receive a loading dose of clopidogrel (≥ 300 mg) and aspirin (≥ 300 mg) if not currently on chronic anti-platelet therapy 24 hrs prior to the index procedure. Patients should remain on 75mg of clopidogrel daily for at least 12 months and on ≥ 75 mg of aspirin indefinitely or at least for the length of the study follow-up period of 5 years.
- All patients will undergo angiography at the 6 month follow-up.
- IVUS and OCT will be conducted at baseline, 6 and 24 and/or 36 months in a subset of the first 35 patients enrolled at select sites. This subset of patients will also undergo angiography at the 24 and/or 36 month follow-up.
- Multislice computed tomography (MSCT) will be conducted will be conducted at 12 months in the subset of the first 35 patients enrolled at select sites.

## **Key Inclusion Criteria**

Patients have a planned intervention of up to two native coronary artery lesions located in separate epicardial territories, one designated the target lesion and the other a non-target lesion, which meet the following criteria:

The non-target lesion must be treated first using a single, approved 'olimus drug eluting stent. If uncomplicated and considered optimal as defined by below, the target lesion can then be treated.

Optimal treatment of non-target lesion:

- a. < 20% residual stenosis by visual assessment
- b. no evidence of dissection
- c. no evidence of thrombus in the target lesion or vessel
- d. TIMI 3 flow

No other restrictions are placed on the non-target lesion. The patient and target lesion must meet all patient inclusion criteria and no exclusion criteria.

Target Lesion inclusion criteria:

- de novo
- The target lesion reference site must be between  $\geq 2.75$  mm and  $\leq 3.5$  mm in diameter assessed by online QCA
- The target vessel must be a major coronary artery or major branch with a visually estimated stenosis of  $\geq 50\%$  and <100% with TIMI flow of  $\geq 1$
- The visually estimated target lesion length is ≤ 10mm or ≤ 14 mm and must be able to be covered by a single 14 mm or 18 mm DESolve® Scaffold
- Percutaneous intervention of lesions in a non-target vessel if:
  - o Not part of a another clinical investigation
  - $\circ$   $\geq$  30 days prior to the study index procedure
  - $\circ$   $\geq$  9 months after the study index procedure (planned)
  - Treatment of a single, non-target lesion located in a separate major epicardial vessel (defined as LAD with septal and diagonal branches, LCX with obtuse marginal and/or ramus intermedius branches and RCA and any of its branches) attempted during the index procedure must be completed first using an approved 'olimus drug eluting stent. If the procedure is deemed uncomplicated and optimal, treatment of the target lesion with the DESolve scaffold can be considered.
- Percutaneous intervention of lesions in the target vessel if:
  - Not part of a clinical investigation
  - $\circ$   $\geq$  6 months prior to the study index procedure
  - $\circ \geq 9$  months after the study index procedure (planned)
  - Previous intervention was distal to and >10mm from the target lesion
- The patient must be an acceptable candidate for coronary artery bypass surgery

### Patients must not have any of the following: **Key Exclusion** Criteria An untreated significant lesion of > 40% diameter stenosis remaining proximal or distal to the target site after the planned intervention The lesion is aorto-ostial in location, an unprotected left main lesion, a lesion within 5 mm of the origin of the LAD or LCX, or involves a major side branch < 2mm in diameter Previous placement of a stent proximal to or within 10 mm of the target lesion Total occlusion or < TIMI 1 coronary flow in the target vessel The proximal target vessel or target lesion contains thrombus, moderate to severe calcification or exhibits severe tortuosity (≥ 45° angulation) by visual assessment High probability that treatment other than PTCA or stenting will be required for treatment of the same lesion Patient is a woman of childbearing potential, pregnant or nursing Patient has received brachytherapy in an epicardial vessel Any use of rotablator at the index procedure The patient was diagnosed with an acute myocardial infarction (AMI) within the past 72 hours and the CK and CKMB have not returned to normal and the patient is experiencing clinical symptoms indicative of ongoing ischemia Analysis Populations in this observational study. **Statistical Analysis** Modified-Intent-to-Treat Evaluable Population The modified-intent-to-treat evaluable population will consist of patients who have received the investigational device at the target lesion, who have no major procedural protocol deviations (e.g. scaffold implanted in a nonnative coronary artery), no bailout scaffolding and for whom follow-up data

is available.

Intent-to-Treat Population

The intent-to-treat population will consist of all patients enrolled in the study, regardless of the treatment actually received for the target lesion.

Statistical Analyses

Detailed descriptive analyses of endpoints will be performed after each follow-up time point. No effort will be made to impute or extrapolate data to replace missing values. All calculations will be based on available data with missing data excluded. Any unused or spurious data will be noted as appropriate in the final report.

All clinical, angiographic, IVUS and OCT endpoints will be analyzed for the modified-intent-to-treat evaluable population. Descriptive statistics will be presented.

For binary variables such as MACE, ABR, TLR, TVF, and persistent incomplete apposition of the scaffold, counts, percentages, and exact 95% confidence intervals using Clopper-Pearson's method will be calculated.

For continuous variables, means, standard deviations, and 95% confidence intervals for the mean using the Gaussian approximation will be calculated. If the assumption of normality seems untenable, nonparametric summary statistics will be presented instead.

For time-to-event variables, such as time to TVF, survival curves will be constructed using Kaplan-Meier estimates.